CLINICAL TRIAL: NCT00821132
Title: Identification of Genes Causing Familial ALS or Increasing Risk for Sporadic ALS and ALS With Frontotemporal Dementia and Understanding Disease Mechanism.
Brief Title: Genetics of Familial and Sporadic ALS
Acronym: ALS
Status: Completed | Type: Observational
Sponsor: Northwestern University (Other)
Responsible Party: Principal Investigator, Teepu Siddique, Director, Division of Neuromuscular Medicine, Northwestern University
Other Study IDs: Lab01; RO1N505641-04 (Other: NINDS)
Record Dates: First submitted 2009-01-09; First posted 2009-01-13 (Estimated); Last update posted 2023-01-26 (Actual); Status verified 2023-01

CONDITIONS: Amyotrophic Lateral Sclerosis (ALS); Familial Amyotrophic Lateral Sclerosis; ALS With Frontotemporal Dementia (ALS/FTD); Lou Gehrig's Disease; Motor Neuron Disease (MND); Primary Lateral Sclerosis (PLS); Sporadic ALS (SALS)
Keywords: FALS; ALS; ALS/FTD; SALS; MND; PLS
MeSH Terms: conditions — Amyotrophic Lateral Sclerosis; Motor Neuron Disease

STUDY DESIGN:
Observational Model: Family Based | Time Perspective: Other
Biospecimen Retention: Samples With DNA — Whole blood and/or skin and cerebrospinal fluid (CSF) samples
  The investigators also collect brain and spinal cord tissue specimens.
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- ALS families: Patients with either inherited or sporadic ALS or PLS and selected family members
  Interventions: Other: Genetic study of ALS families

INTERVENTIONS:
Other: Genetic study of ALS families — Collection and analysis of genetic material, medical and family histories from families with ALS
  Other Names: familial ALS; sporadic ALS; genetics of ALS; ALS with frontotemporal dementia; Motor Neuron Disease; Lou Gehrig's disease; neuromuscular disease; Frontotemporal dementia; Primary Lateral Sclerosis; Amyotrophic lateral sclerosis

SUMMARY:
We are collecting blood samples, clinical and family information from ALS (amyotrophic lateral sclerosis) patients and their families to identify causes of ALS and ALS/dementia.

DETAILED DESCRIPTION:
The investigators' long term goals are to improve diagnosis and develop effective treatments that arrest or ameliorate symptoms of ALS, and possibly delay or prevent disease onset in individuals at risk for developing familial ALS (FALS). In order to do this one must understand how disease develops at a molecular level. Identification of genes that increase risk for developing all types of ALS will reveal the pathways of molecular events that are involved in ALS.

The investigators are collecting blood samples, family and medical histories of patients with all types of ALS, (familial and sporadic, with and without frontotemporal dementia, and primary lateral sclerosis and particular family members. Samples are coded to maintain confidentiality. Travel is not necessary.

As well as seeking to identify new genes implicated in ALS, the investigators continue our study of families with known genetic mutations to more fully characterize that disease mechanism.

Linkage analysis and affected relative pair analysis will be used to identify causative FALS genes and disequilibrium analysis and association studies are being done for sporadic ALS.

Results from these studies will provide insight into the underlying disease mechanisms of ALS and provide targets for therapeutic interventions.

ELIGIBILITY:
Inclusion Criteria:

* Patients with Amyotrophic Lateral Sclerosis or ALS and frontotemporal dementia
* Selected family members, generally brothers and sisters of an ALS patient, the patient's parents

Exclusion Criteria:

* Under 18 years old

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Open to all ALS patients and selected family members
Sampling Method: Non-Probability Sample
Enrollment: 13521 (Actual)
Dates: Start 1991-01 (Actual); Primary Completion 2023-01 (Actual); Study Completion 2023-01 (Actual)

PRIMARY OUTCOMES:
Identification of genes that increase risk for sporadic ALS or cause inherited ALS. | Dec 2025
  Study of each identified gene will help us understand the molecular events that produce different types of ALS. This will aid in identification of markers that may be associated with each type which will assist with diagnosis and may provide targets for rational therapy.

CONTACTS AND LOCATIONS:
Overall Officials: Teepu Siddique, MD, Principal Investigator — Northwestern University Feinberg School of Medicine
Locations (1):
- Northwestern University Feinberg School of Medicine, Chicago, Illinois, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Pytte J, Anderton RS, Flynn LL, Theunissen F, Jiang L, Pitout I, James I, Mastaglia FL, Saunders AM, Bedlack R, Siddique T, Siddique N, Akkari PA. Association of a structural variant within the SQSTM1 gene with amyotrophic lateral sclerosis. Neurol Genet. 2020 Feb 27;6(2):e406. doi: 10.1212/NXG.0000000000000406. eCollection 2020 Apr. PMID 32185242
- [Background] Deng HX, Zhai H, Shi Y, Liu G, Lowry J, Liu B, Ryan EB, Yan J, Yang Y, Zhang N, Yang Z, Liu E, Ma YC, Siddique T. Efficacy and long-term safety of CRISPR/Cas9 genome editing in the SOD1-linked mouse models of ALS. Commun Biol. 2021 Mar 25;4(1):396. doi: 10.1038/s42003-021-01942-4. PMID 33767386
- [Background] Ryan EB, Yan J, Miller N, Dayanidhi S, Ma YC, Deng HX, Siddique T. Early death of ALS-linked CHCHD10-R15L transgenic mice with central nervous system, skeletal muscle, and cardiac pathology. iScience. 2021 Jan 18;24(2):102061. doi: 10.1016/j.isci.2021.102061. eCollection 2021 Feb 19. PMID 33659869
- [Background] Ryan EB, Deng HX. Does Somatic Mosaicism Account for Some Sporadic ALS? Neurol Genet. 2021 Jan 12;7(1):e555. doi: 10.1212/NXG.0000000000000555. eCollection 2021 Feb. No abstract available. PMID 33977141
- [Background] Lowry JL, Ryan EB, Esengul YT, Siddique N, Siddique T. Intricacies of aetiology in intrafamilial degenerative disease. Brain Commun. 2020 Oct 6;2(2):fcaa120. doi: 10.1093/braincomms/fcaa120. eCollection 2020. PMID 33134917
- [Background] Ortega JA, Daley EL, Kour S, Samani M, Tellez L, Smith HS, Hall EA, Esengul YT, Tsai YH, Gendron TF, Donnelly CJ, Siddique T, Savas JN, Pandey UB, Kiskinis E. Nucleocytoplasmic Proteomic Analysis Uncovers eRF1 and Nonsense-Mediated Decay as Modifiers of ALS/FTD C9orf72 Toxicity. Neuron. 2020 Apr 8;106(1):90-107.e13. doi: 10.1016/j.neuron.2020.01.020. Epub 2020 Feb 13. PMID 32059759
- [Background] Wu JJ, Cai A, Greenslade JE, Higgins NR, Fan C, Le NTT, Tatman M, Whiteley AM, Prado MA, Dieriks BV, Curtis MA, Shaw CE, Siddique T, Faull RLM, Scotter EL, Finley D, Monteiro MJ. ALS/FTD mutations in UBQLN2 impede autophagy by reducing autophagosome acidification through loss of function. Proc Natl Acad Sci U S A. 2020 Jun 30;117(26):15230-15241. doi: 10.1073/pnas.1917371117. Epub 2020 Jun 8. PMID 32513711
- [Background] Silani V, Corcia P, Harms MB, Rouleau G, Siddique T, Ticozzi N. Genetics of primary lateral sclerosis. Amyotroph Lateral Scler Frontotemporal Degener. 2020 Nov;21(sup1):28-34. doi: 10.1080/21678421.2020.1837177. PMID 33602012
- [Background] Edens BM, Yan J, Miller N, Deng HX, Siddique T, Ma YC. A novel ALS-associated variant in UBQLN4 regulates motor axon morphogenesis. Elife. 2017 May 2;6:e25453. doi: 10.7554/eLife.25453. PMID 28463112
- [Result] Rosen DR, Siddique T, Patterson D, Figlewicz DA, Sapp P, Hentati A, Donaldson D, Goto J, O'Regan JP, Deng HX, et al. Mutations in Cu/Zn superoxide dismutase gene are associated with familial amyotrophic lateral sclerosis. Nature. 1993 Mar 4;362(6415):59-62. doi: 10.1038/362059a0. PMID 8446170
- [Result] Chen W, Saeed M, Mao H, Siddique N, Dellefave L, Hung WY, Deng HX, Sufit RL, Heller SL, Haines JL, Pericak-Vance M, Siddique T. Lack of association of VEGF promoter polymorphisms with sporadic ALS. Neurology. 2006 Aug 8;67(3):508-10. doi: 10.1212/01.wnl.0000227926.42370.04. PMID 16894118
- [Result] Li YJ, Pericak-Vance MA, Haines JL, Siddique N, McKenna-Yasek D, Hung WY, Sapp P, Allen CI, Chen W, Hosler B, Saunders AM, Dellefave LM, Brown RH, Siddique T. Apolipoprotein E is associated with age at onset of amyotrophic lateral sclerosis. Neurogenetics. 2004 Dec;5(4):209-13. doi: 10.1007/s10048-004-0193-0. Epub 2004 Oct 2. PMID 15657798
- [Result] Yang Y, Hentati A, Deng HX, Dabbagh O, Sasaki T, Hirano M, Hung WY, Ouahchi K, Yan J, Azim AC, Cole N, Gascon G, Yagmour A, Ben-Hamida M, Pericak-Vance M, Hentati F, Siddique T. The gene encoding alsin, a protein with three guanine-nucleotide exchange factor domains, is mutated in a form of recessive amyotrophic lateral sclerosis. Nat Genet. 2001 Oct;29(2):160-5. doi: 10.1038/ng1001-160. PMID 11586297
- [Result] Hentati A, Ouahchi K, Pericak-Vance MA, Nijhawan D, Ahmad A, Yang Y, Rimmler J, Hung W, Schlotter B, Ahmed A, Ben Hamida M, Hentati F, Siddique T. Linkage of a commoner form of recessive amyotrophic lateral sclerosis to chromosome 15q15-q22 markers. Neurogenetics. 1998 Dec;2(1):55-60. doi: 10.1007/s100480050052. PMID 9933301
- [Result] Ajroud-Driss S, Saeed M, Khan H, Siddique N, Hung WY, Sufit R, Heller S, Armstrong J, Casey P, Siddique T, Lukas TJ. Riluzole metabolism and CYP1A1/2 polymorphisms in patients with ALS. Amyotroph Lateral Scler. 2007 Oct;8(5):305-9. doi: 10.1080/17482960701500650. PMID 17852022
- [Result] Deng HX, Shi Y, Furukawa Y, Zhai H, Fu R, Liu E, Gorrie GH, Khan MS, Hung WY, Bigio EH, Lukas T, Dal Canto MC, O'Halloran TV, Siddique T. Conversion to the amyotrophic lateral sclerosis phenotype is associated with intermolecular linked insoluble aggregates of SOD1 in mitochondria. Proc Natl Acad Sci U S A. 2006 May 2;103(18):7142-7. doi: 10.1073/pnas.0602046103. Epub 2006 Apr 24. PMID 16636275
- [Result] Saeed M, Siddique N, Hung WY, Usacheva E, Liu E, Sufit RL, Heller SL, Haines JL, Pericak-Vance M, Siddique T. Paraoxonase cluster polymorphisms are associated with sporadic ALS. Neurology. 2006 Sep 12;67(5):771-6. doi: 10.1212/01.wnl.0000227187.52002.88. Epub 2006 Jul 5. PMID 16822964
- [Result] Hosler BA, Siddique T, Sapp PC, Sailor W, Huang MC, Hossain A, Daube JR, Nance M, Fan C, Kaplan J, Hung WY, McKenna-Yasek D, Haines JL, Pericak-Vance MA, Horvitz HR, Brown RH Jr. Linkage of familial amyotrophic lateral sclerosis with frontotemporal dementia to chromosome 9q21-q22. JAMA. 2000 Oct 4;284(13):1664-9. doi: 10.1001/jama.284.13.1664. PMID 11015796
- [Result] Yan J, Deng HX, Siddique N, Fecto F, Chen W, Yang Y, Liu E, Donkervoort S, Zheng JG, Shi Y, Ahmeti KB, Brooks B, Engel WK, Siddique T. Frameshift and novel mutations in FUS in familial amyotrophic lateral sclerosis and ALS/dementia. Neurology. 2010 Aug 31;75(9):807-14. doi: 10.1212/WNL.0b013e3181f07e0c. Epub 2010 Jul 28. PMID 20668259
- [Result] Deng HX, Zhai H, Bigio EH, Yan J, Fecto F, Ajroud K, Mishra M, Ajroud-Driss S, Heller S, Sufit R, Siddique N, Mugnaini E, Siddique T. FUS-immunoreactive inclusions are a common feature in sporadic and non-SOD1 familial amyotrophic lateral sclerosis. Ann Neurol. 2010 Jun;67(6):739-48. doi: 10.1002/ana.22051. PMID 20517935
- [Result] Zhou J, Yi J, Fu R, Liu E, Siddique T, Rios E, Deng HX. Hyperactive intracellular calcium signaling associated with localized mitochondrial defects in skeletal muscle of an animal model of amyotrophic lateral sclerosis. J Biol Chem. 2010 Jan 1;285(1):705-12. doi: 10.1074/jbc.M109.041319. Epub 2009 Nov 4. PMID 19889637
- [Result] Kwiatkowski TJ Jr, Bosco DA, Leclerc AL, Tamrazian E, Vanderburg CR, Russ C, Davis A, Gilchrist J, Kasarskis EJ, Munsat T, Valdmanis P, Rouleau GA, Hosler BA, Cortelli P, de Jong PJ, Yoshinaga Y, Haines JL, Pericak-Vance MA, Yan J, Ticozzi N, Siddique T, McKenna-Yasek D, Sapp PC, Horvitz HR, Landers JE, Brown RH Jr. Mutations in the FUS/TLS gene on chromosome 16 cause familial amyotrophic lateral sclerosis. Science. 2009 Feb 27;323(5918):1205-8. doi: 10.1126/science.1166066. PMID 19251627
- [Result] Wang L, Deng HX, Grisotti G, Zhai H, Siddique T, Roos RP. Wild-type SOD1 overexpression accelerates disease onset of a G85R SOD1 mouse. Hum Mol Genet. 2009 May 1;18(9):1642-51. doi: 10.1093/hmg/ddp085. Epub 2009 Feb 19. PMID 19233858
- [Result] Saeed M, Yang Y, Deng HX, Hung WY, Siddique N, Dellefave L, Gellera C, Andersen PM, Siddique T. Age and founder effect of SOD1 A4V mutation causing ALS. Neurology. 2009 May 12;72(19):1634-9. doi: 10.1212/01.wnl.0000343509.76828.2a. Epub 2009 Jan 28. PMID 19176896
- [Result] Frutiger K, Lukas TJ, Gorrie G, Ajroud-Driss S, Siddique T. Gender difference in levels of Cu/Zn superoxide dismutase (SOD1) in cerebrospinal fluid of patients with amyotrophic lateral sclerosis. Amyotroph Lateral Scler. 2008 Jun;9(3):184-7. doi: 10.1080/17482960801984358. PMID 18574763
- [Result] Deng HX, Jiang H, Fu R, Zhai H, Shi Y, Liu E, Hirano M, Dal Canto MC, Siddique T. Molecular dissection of ALS-associated toxicity of SOD1 in transgenic mice using an exon-fusion approach. Hum Mol Genet. 2008 Aug 1;17(15):2310-9. doi: 10.1093/hmg/ddn131. Epub 2008 Apr 18. PMID 18424447
- [Result] Deng HX, Chen W, Hong ST, Boycott KM, Gorrie GH, Siddique N, Yang Y, Fecto F, Shi Y, Zhai H, Jiang H, Hirano M, Rampersaud E, Jansen GH, Donkervoort S, Bigio EH, Brooks BR, Ajroud K, Sufit RL, Haines JL, Mugnaini E, Pericak-Vance MA, Siddique T. Mutations in UBQLN2 cause dominant X-linked juvenile and adult-onset ALS and ALS/dementia. Nature. 2011 Aug 21;477(7363):211-5. doi: 10.1038/nature10353. PMID 21857683
- [Result] Deng HX, Klein CJ, Yan J, Shi Y, Wu Y, Fecto F, Yau HJ, Yang Y, Zhai H, Siddique N, Hedley-Whyte ET, Delong R, Martina M, Dyck PJ, Siddique T. Scapuloperoneal spinal muscular atrophy and CMT2C are allelic disorders caused by alterations in TRPV4. Nat Genet. 2010 Feb;42(2):165-9. doi: 10.1038/ng.509. Epub 2009 Dec 27. PMID 20037587
- [Result] Fecto F, Yan J, Vemula SP, Liu E, Yang Y, Chen W, Zheng JG, Shi Y, Siddique N, Arrat H, Donkervoort S, Ajroud-Driss S, Sufit RL, Heller SL, Deng HX, Siddique T. SQSTM1 mutations in familial and sporadic amyotrophic lateral sclerosis. Arch Neurol. 2011 Nov;68(11):1440-6. doi: 10.1001/archneurol.2011.250. PMID 22084127
- [Result] Bigio EH, Wu JY, Deng HX, Bit-Ivan EN, Mao Q, Ganti R, Peterson M, Siddique N, Geula C, Siddique T, Mesulam M. Inclusions in frontotemporal lobar degeneration with TDP-43 proteinopathy (FTLD-TDP) and amyotrophic lateral sclerosis (ALS), but not FTLD with FUS proteinopathy (FTLD-FUS), have properties of amyloid. Acta Neuropathol. 2013 Mar;125(3):463-5. doi: 10.1007/s00401-013-1089-6. Epub 2013 Feb 3. No abstract available. PMID 23378033
- [Result] Ahmeti KB, Ajroud-Driss S, Al-Chalabi A, Andersen PM, Armstrong J, Birve A, Blauw HM, Brown RH, Bruijn L, Chen W, Chio A, Comeau MC, Cronin S, Diekstra FP, Soraya Gkazi A, Glass JD, Grab JD, Groen EJ, Haines JL, Hardiman O, Heller S, Huang J, Hung WY; ITALSGEN consortium; Jaworski JM, Jones A, Khan H, Landers JE, Langefeld CD, Leigh PN, Marion MC, McLaughlin RL, Meininger V, Melki J, Miller JW, Mora G, Pericak-Vance MA, Rampersaud E, Robberecht W, Russell LP, Salachas F, Saris CG, Shatunov A, Shaw CE, Siddique N, Siddique T, Smith BN, Sufit R, Topp S, Traynor BJ, Vance C, van Damme P, van den Berg LH, van Es MA, van Vught PW, Veldink JH, Yang Y, Zheng JG; ALSGEN Consortium. Age of onset of amyotrophic lateral sclerosis is modulated by a locus on 1p34.1. Neurobiol Aging. 2013 Jan;34(1):357.e7-19. doi: 10.1016/j.neurobiolaging.2012.07.017. Epub 2012 Sep 5. PMID 22959728
- [Result] Kwan JY, Jeong SY, Van Gelderen P, Deng HX, Quezado MM, Danielian LE, Butman JA, Chen L, Bayat E, Russell J, Siddique T, Duyn JH, Rouault TA, Floeter MK. Iron accumulation in deep cortical layers accounts for MRI signal abnormalities in ALS: correlating 7 tesla MRI and pathology. PLoS One. 2012;7(4):e35241. doi: 10.1371/journal.pone.0035241. Epub 2012 Apr 17. PMID 22529995
- [Result] Fecto F, Siddique T. SIGMAR1 mutations, genetic heterogeneity at the chromosome 9p locus, and the expanding etiological diversity of amyotrophic lateral sclerosis. Ann Neurol. 2011 Dec;70(6):867-70. doi: 10.1002/ana.22648. No abstract available. PMID 22190360
- [Result] Fecto F, Siddique T. What is repeated in ALS and FTLD. Lancet Neurol. 2012 Jan;11(1):25-7. doi: 10.1016/S1474-4422(11)70275-7. Epub 2011 Dec 7. No abstract available. PMID 22154784
- [Result] Siddique T, Ajroud-Driss S. Familial amyotrophic lateral sclerosis, a historical perspective. Acta Myol. 2011 Oct;30(2):117-20. PMID 22106714
- [Result] Deng HX, Bigio EH, Siddique T. Detection of protein aggregation in neurodegenerative diseases. Methods Mol Biol. 2011;793:259-72. doi: 10.1007/978-1-61779-328-8_17. PMID 21913106
- [Result] Fecto F, Siddique T. Making connections: pathology and genetics link amyotrophic lateral sclerosis with frontotemporal lobe dementia. J Mol Neurosci. 2011 Nov;45(3):663-75. doi: 10.1007/s12031-011-9637-9. Epub 2011 Sep 7. PMID 21901496
- [Result] Deng HX, Bigio EH, Zhai H, Fecto F, Ajroud K, Shi Y, Yan J, Mishra M, Ajroud-Driss S, Heller S, Sufit R, Siddique N, Mugnaini E, Siddique T. Differential involvement of optineurin in amyotrophic lateral sclerosis with or without SOD1 mutations. Arch Neurol. 2011 Aug;68(8):1057-61. doi: 10.1001/archneurol.2011.178. PMID 21825243
- [Result] Subramony SH, Ashizawa T, Langford L, McKenna R, Avvaru B, Siddique T, Vedanarayanan V. Confirmation of the severe phenotypic effect of serine at codon 41 of the superoxide dismutase 1 gene. Muscle Nerve. 2011 Oct;44(4):499-502. doi: 10.1002/mus.22117. Epub 2011 Jul 13. PMID 21755517
- [Result] Fecto F, Shi Y, Huda R, Martina M, Siddique T, Deng HX. Mutant TRPV4-mediated toxicity is linked to increased constitutive function in axonal neuropathies. J Biol Chem. 2011 May 13;286(19):17281-91. doi: 10.1074/jbc.M111.237685. Epub 2011 Mar 21. PMID 21454511
- [Result] Yasser S, Fecto F, Siddique T, Sheikh KA, Athar P. An unusual case of familial ALS and cerebellar ataxia. Amyotroph Lateral Scler. 2010 Dec;11(6):568-70. doi: 10.3109/17482961003636874. Epub 2010 Jun 14. PMID 20540686
- [Result] Siddique N, Siddique T. Amyotrophic Lateral Sclerosis Overview. 2001 Mar 23 [updated 2023 Sep 28]. In: Adam MP, Bick S, Mirzaa GM, Pagon RA, Wallace SE, Amemiya A, editors. GeneReviews(R) [Internet]. Seattle (WA): University of Washington, Seattle; 1993-2026. Available from http://www.ncbi.nlm.nih.gov/books/NBK1450/ PMID 20301623
- [Result] Fogh I, Ratti A, Gellera C, Lin K, Tiloca C, Moskvina V, Corrado L, Soraru G, Cereda C, Corti S, Gentilini D, Calini D, Castellotti B, Mazzini L, Querin G, Gagliardi S, Del Bo R, Conforti FL, Siciliano G, Inghilleri M, Sacca F, Bongioanni P, Penco S, Corbo M, Sorbi S, Filosto M, Ferlini A, Di Blasio AM, Signorini S, Shatunov A, Jones A, Shaw PJ, Morrison KE, Farmer AE, Van Damme P, Robberecht W, Chio A, Traynor BJ, Sendtner M, Melki J, Meininger V, Hardiman O, Andersen PM, Leigh NP, Glass JD, Overste D, Diekstra FP, Veldink JH, van Es MA, Shaw CE, Weale ME, Lewis CM, Williams J, Brown RH, Landers JE, Ticozzi N, Ceroni M, Pegoraro E, Comi GP, D'Alfonso S, van den Berg LH, Taroni F, Al-Chalabi A, Powell J, Silani V; SLAGEN Consortium and Collaborators. A genome-wide association meta-analysis identifies a novel locus at 17q11.2 associated with sporadic amyotrophic lateral sclerosis. Hum Mol Genet. 2014 Apr 15;23(8):2220-31. doi: 10.1093/hmg/ddt587. Epub 2013 Nov 20. PMID 24256812
- [Result] Wang X, Blanchard J, Grundke-Iqbal I, Wegiel J, Deng HX, Siddique T, Iqbal K. Alzheimer disease and amyotrophic lateral sclerosis: an etiopathogenic connection. Acta Neuropathol. 2014 Feb;127(2):243-56. doi: 10.1007/s00401-013-1175-9. Epub 2013 Oct 18. PMID 24136402
- [Result] Fecto F, Siddique T. UBQLN2/P62 cellular recycling pathways in amyotrophic lateral sclerosis and frontotemporal dementia. Muscle Nerve. 2012 Feb;45(2):157-62. doi: 10.1002/mus.23278. PMID 22246868
- [Result] Gallardo G, Barowski J, Ravits J, Siddique T, Lingrel JB, Robertson J, Steen H, Bonni A. An alpha2-Na/K ATPase/alpha-adducin complex in astrocytes triggers non-cell autonomous neurodegeneration. Nat Neurosci. 2014 Dec;17(12):1710-9. doi: 10.1038/nn.3853. Epub 2014 Oct 26. PMID 25344630
- [Result] Fawzi AA, Simonett JM, Purta P, Moss HE, Lowry JL, Deng HX, Siddique N, Sufit R, Bigio EH, Volpe NJ, Siddique T. Clinicopathologic report of ocular involvement in ALS patients with C9orf72 mutation. Amyotroph Lateral Scler Frontotemporal Degener. 2014 Dec;15(7-8):569-80. doi: 10.3109/21678421.2014.951941. Epub 2014 Oct 16. PMID 25319030
- [Result] Gorrie GH, Fecto F, Radzicki D, Weiss C, Shi Y, Dong H, Zhai H, Fu R, Liu E, Li S, Arrat H, Bigio EH, Disterhoft JF, Martina M, Mugnaini E, Siddique T, Deng HX. Dendritic spinopathy in transgenic mice expressing ALS/dementia-linked mutant UBQLN2. Proc Natl Acad Sci U S A. 2014 Oct 7;111(40):14524-9. doi: 10.1073/pnas.1405741111. Epub 2014 Sep 22. PMID 25246588
- [Result] Hartzfeld DE, Siddique N, Victorson D, O'Neill S, Kinsley L, Siddique T. Reproductive decision-making among individuals at risk for familial amyotrophic lateral sclerosis. Amyotroph Lateral Scler Frontotemporal Degener. 2015 Mar;16(1-2):114-9. doi: 10.3109/21678421.2014.951945. Epub 2014 Sep 10. PMID 25204983
- [Result] Ajroud-Driss S, Siddique T. Sporadic and hereditary amyotrophic lateral sclerosis (ALS). Biochim Biophys Acta. 2015 Apr;1852(4):679-84. doi: 10.1016/j.bbadis.2014.08.010. Epub 2014 Sep 1. PMID 25193032
- [Result] Fecto F, Esengul YT, Siddique T. Protein recycling pathways in neurodegenerative diseases. Alzheimers Res Ther. 2014 Mar 6;6(2):13. doi: 10.1186/alzrt243. eCollection 2014. PMID 25031631
- [Result] Lukas TJ, Schiltz GE, Arrat H, Scheidt K, Siddique T. Discovery of 1,3,4-oxidiazole scaffold compounds as inhibitors of superoxide dismutase expression. Bioorg Med Chem Lett. 2014 Mar 15;24(6):1532-7. doi: 10.1016/j.bmcl.2014.01.078. Epub 2014 Feb 8. PMID 24560539
- [Result] Al-Chalabi A, Kwak S, Mehler M, Rouleau G, Siddique T, Strong M, Leigh PN. Genetic and epigenetic studies of amyotrophic lateral sclerosis. Amyotroph Lateral Scler Frontotemporal Degener. 2013 May;14 Suppl 1:44-52. doi: 10.3109/21678421.2013.778571. PMID 23678879
- [Result] Volpe NJ, Simonett J, Fawzi AA, Siddique T. Ophthalmic Manifestations of Amyotrophic Lateral Sclerosis (An American Ophthalmological Society Thesis). Trans Am Ophthalmol Soc. 2015;113:T12. PMID 26877563
- [Result] Arrat H, Lukas TJ, Siddique T. ACTH (Acthar Gel) Reduces Toxic SOD1 Protein Linked to Amyotrophic Lateral Sclerosis in Transgenic Mice: A Novel Observation. PLoS One. 2015 May 8;10(5):e0125638. doi: 10.1371/journal.pone.0125638. eCollection 2015. PMID 25955410
- [Result] Radzicki D, Liu E, Deng HX, Siddique T, Martina M. Early Impairment of Synaptic and Intrinsic Excitability in Mice Expressing ALS/Dementia-Linked Mutant UBQLN2. Front Cell Neurosci. 2016 Sep 20;10:216. doi: 10.3389/fncel.2016.00216. eCollection 2016. PMID 27703430
- [Result] Yang Y, Zhang L, Lynch DR, Lukas T, Ahmeti K, Sleiman PM, Ryan E, Schadt KA, Newman JH, Deng HX, Siddique N, Siddique T. Compound heterozygote mutations in SPG7 in a family with adult-onset primary lateral sclerosis. Neurol Genet. 2016 Mar 3;2(2):e60. doi: 10.1212/NXG.0000000000000060. eCollection 2016 Apr. PMID 27123479
- [Result] Simonett JM, Huang R, Siddique N, Farsiu S, Siddique T, Volpe NJ, Fawzi AA. Macular sub-layer thinning and association with pulmonary function tests in Amyotrophic Lateral Sclerosis. Sci Rep. 2016 Jul 7;6:29187. doi: 10.1038/srep29187. PMID 27383525
- [Result] Lee S, Shang Y, Redmond SA, Urisman A, Tang AA, Li KH, Burlingame AL, Pak RA, Jovicic A, Gitler AD, Wang J, Gray NS, Seeley WW, Siddique T, Bigio EH, Lee VM, Trojanowski JQ, Chan JR, Huang EJ. Activation of HIPK2 Promotes ER Stress-Mediated Neurodegeneration in Amyotrophic Lateral Sclerosis. Neuron. 2016 Jul 6;91(1):41-55. doi: 10.1016/j.neuron.2016.05.021. Epub 2016 Jun 16. PMID 27321923
- [Result] Deng HX, Shi Y, Yang Y, Ahmeti KB, Miller N, Huang C, Cheng L, Zhai H, Deng S, Nuytemans K, Corbett NJ, Kim MJ, Deng H, Tang B, Yang Z, Xu Y, Chan P, Huang B, Gao XP, Song Z, Liu Z, Fecto F, Siddique N, Foroud T, Jankovic J, Ghetti B, Nicholson DA, Krainc D, Melen O, Vance JM, Pericak-Vance MA, Ma YC, Rajput AH, Siddique T. Identification of TMEM230 mutations in familial Parkinson's disease. Nat Genet. 2016 Jul;48(7):733-9. doi: 10.1038/ng.3589. Epub 2016 Jun 6. PMID 27270108
- [Result] Bali T, Self W, Liu J, Siddique T, Wang LH, Bird TD, Ratti E, Atassi N, Boylan KB, Glass JD, Maragakis NJ, Caress JB, McCluskey LF, Appel SH, Wymer JP, Gibson S, Zinman L, Mozaffar T, Callaghan B, McVey AL, Jockel-Balsarotti J, Allred P, Fisher ER, Lopate G, Pestronk A, Cudkowicz ME, Miller TM. Defining SOD1 ALS natural history to guide therapeutic clinical trial design. J Neurol Neurosurg Psychiatry. 2017 Feb;88(2):99-105. doi: 10.1136/jnnp-2016-313521. Epub 2016 Jun 3. PMID 27261500
- [Result] Pytte J, Flynn LL, Anderton RS, Mastaglia FL, Theunissen F, James I, Pfaff A, Koks S, Saunders AM, Bedlack R, Burns DK, Lutz MW, Siddique N, Siddique T, Roses AD, Akkari PA. Disease-modifying effects of an SCAF4 structural variant in a predominantly SOD1 ALS cohort. Neurol Genet. 2020 Jul 1;6(4):e470. doi: 10.1212/NXG.0000000000000470. eCollection 2020 Aug. PMID 32754644